CLINICAL TRIAL: NCT02857686
Title: Forearm Tourniquet With Small Dose Intravenous Lidocaine as a Substitute to Conventional Intravenous Regional Anaesthesia
Brief Title: Forearm Tourniquet With Small Dose Intravenous Lidocaine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer in anesthesia department Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mini IVRA
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Local Anaesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm intravenous regional anesthesia (Active Comparator): tourniquet over the arm and intravenous lidocaine with a dose of 4 mg/kg
  Interventions: Procedure: intravenous regional anaesthesia
- forearm intravenous regional anesthesia (Experimental): tourniquet over the forearm and lidocaine with a dose of 1.5 mg/ kg
  Interventions: Procedure: forearm IVRA

INTERVENTIONS:
Procedure: intravenous regional anaesthesia — tourniquet over the arm and intravenous lidocaine with a dose of 4 mg/kg
  Arms: arm intravenous regional anesthesia
Procedure: forearm IVRA — tourniquet over the forearm and lidocaine with a dose of 1.5 mg/ kg
  Arms: forearm intravenous regional anesthesia

SUMMARY:
The safety and effectiveness of the "mini-dose" Bier block, a technique of i.v. regional anesthesia using low-dose lidocaine (1.5 mg/kg) without routine premedication, was evaluated in the emergency department treatment of pediatric upper extremity fractures and dislocations.

DETAILED DESCRIPTION:
this study aimed at comparing IVRA with small dose lidocaine and forearm tourniquet with conventional IVRA with arm tourniquet and usual lidocaine dose

ELIGIBILITY:
Inclusion Criteria:

* ASA(American society of anesthesia) I, II , consent, forearm or arm surgery

Exclusion Criteria:

* ASA(American society of anesthesia) III or more, allergy, refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
pain | 2 hours
  visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided